CLINICAL TRIAL: NCT05154279
Title: The Effect of Intramyometrial Injection of Terlipressin Versus Intramyometrial Injection of Carbitocin on Hemoglobin and Blood Loss During Laparoscopic Myomectomy Operations: Double Blinded Randomized Placebo-Controlled Trial
Brief Title: The Effect of Intramyometrial Injection of Terlipressin Versus Intramyometrial Injection of Carbitocin on Hemoglobin and Blood Loss During Laparoscopic Myomectomy Operations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Elbanna Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Elbanna_005
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-10

CONDITIONS: Laparoscopic Myomectomy
Keywords: laparoscopic myomectomy; Terlipressin; carbitocin
MeSH Terms: interventions — Terlipressin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- intramyometrial Terlipressin (Active Comparator): intramyometrial injection of Terlipressin in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin
- intramyometrial carbitocin (Active Comparator): intramyometrial injection of Carbetocin in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin
- intramyometrial saline (Placebo Comparator): intramyometrial injection of saline in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — intramyometrial terlipressin vs carbitocin vs saline as placebo
  Other Names: carbitocin; saline

SUMMARY:
Our study aims to evaluate the efficacy of intramyometrial injection of Terlipressin versus intramyometrial injection of Carbetocin on hemoglobin level in women undergoing abdominal myomectomy. Moreover, to evaluate their efficacy in decreasing blood loss on operative time and to describe the injection sequelae for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

DETAILED DESCRIPTION:
Fibroids are firm benign tumors that are made of smooth muscle cells and fibrous connective tissue. Benign uterine leiomyomas (fibroids) are the most common pelvic tumor in women, affecting 20-40% of all women over the age of 35 and 50% of African American women. Approximately 20-40% of women with fibroids experience significant symptoms and consult gynecologic care. However, their true prevalence is probably underestimated . The most common clinical symptoms include abnormal uterine bleeding, dysmenorrhea, pelvic pain, infertility, and recurrent pregnancy loss . Less commonly, women with a uterine mass presumed to be a leiomyoma are found to have a uterine sarcoma or a leiomyoma variant Although hysterectomy is the definitive treatment for myomas, myomectomy remains the gold-standard treatment for women wishing to preserve their uterus and fertility . However, bleeding is often a problem in a myomectomy and can result in intra-operative hypovolaemic shock, post-operative anemia, and delayed recovery .

Three common causes of increased blood loss during abdominal myomectomy are poor surgical technique, the complexity of intra-abdominal pathology (such as low corpus, intra- ligamentous myomas, or obliteration of culde-sac), and the excessive loss of intrauterine blood during dissection of the myomas .

The current treatments for uterine fibroids are many, medical as progesterone's and progesterone antagonist's, surgical, and recent myoma therapies as uterine artery embolization, but surgical resection is still the main treatment, including hysterectomy and myomectomy. With hysterectomy, uterine fibroids can be completely cured, but it cannot keep women's reproductive functions. Despite the rate of relapse, myomectomy is still the most popular surgical treatment for fibroids in women .

A myomectomy excises the fibroid(s) and repairs any defect in the uterine wall, while preserving the uterus. For this reason, myomectomy is an option for women who desire future pregnancies or who wish to retain their uterus. After myomectomy, fibroids could recur, which could lead to subsequent intervention(s) . A laparoscope can be used to remove the fibroid(s) through small incisions in the abdominal wall (laparoscopic) or a hysteroscope can be used to reach the fibroid(s) through the cervix (hysteroscopic).

Although laparoscopic myomectomy has been performed since Semm and colleagues described the procedure in late 1970s , the role of laparoscopic myomectomy as a treatment option for symptomatic uterine fibroids has been questioned. Many fibroids that can be easily removed laparoscopically may not require surgical intervention .

Laparoscopic myomectomy was given lukewarm support in the May 2000 American College of Obstetricians and Gynecologists (ACOG) guidelines : The two major concerns with laparoscopic myomectomy versus hysterectomy are the removal of large myomas through small abdominal incisions and the repair of the uterus. The introduction of more efficient morcellators has made the removal easier, although skilled operative technique is necessary because injury to other organs is possible .

Although there are multiple techniques available for laparoscopic suturing, there is controversy as to whether the closure techniques available are equal to those achieved at laparotomy. This is most relevant to women contemplating a future pregnancy. In spite of these reservations, recently published studies indicate that laparoscopic myomectomy may be an appropriate alternative to abdominal myomectomy in well selected patients. Many reproductive surgeons have the prerequisite skills to perform laparoscopic myomectomy, and advances in instruments and techniques have made this approach more accessible to physicians and patients .

Cosmetic consideration and postoperative recovery is always a concern, which results in the request of minimally invasive procedures . Following the initial application of laparoscopic myomectomy (LM) in 1979 by Semm , this minimally invasive technique has become more and more popular worldwide. Conventionally, a three- to four-port wound technique is applied for LM. The main trocar (10 mm port) is inserted through the umbilicus to introduce the video system after pneumoperitoneum insufflation with carbon dioxide. Other two- or three-accessory trocars (5mm port or 10mm port) were inserted into the abdomen over the left lower quadrant, right lower quadrant, and suprapubic area, for the operative instruments and the suction irrigator machine .

As hemorrhage is the main complication so, reduction of intra-operative bleeding has become a major concern. This can be achieved by the use of mechanical or pharmacologic methods, which can be done pre-operative and intra-operative. Mechanical methods include the use of tourniquets and clamps that occlude the uterine blood supply to reduce blood loss during myomectomy. Pharmacologic methods include local Oxytocin injection, vasoconstrictors like Vasopressin .

Pre-operative uterine artery embolization decreases blood loss during myomectomy, but this technique is restricted to particular hospital centers and can be complicated . Laparoscopic uterine artery occlusion has been described as a treatment for symptomatic myomas .

Carbetocin is an Oxytocin derivative exerting effect via the same molecular mechanisms as Oxytocin. It was first described in 1987 and is a long-acting synthetic analog of Oxytocin, with agonist action. The clinical and pharmacological properties of Carbetocin are similar to those of naturally occurring Oxytocin. Its intravenous half-life is 85 to 100 min which is 10 times longer than that of oxytocin. It has a rapid onset and long-lasting action .

Carbetocin and uterine oxytocin receptors in the uterus caused rhythmic contraction, which can increase the frequency of existing contractions as well as uterine tone. During surgery, the uterine smooth muscles were made to contract so that the tumor protrudes from the uterine surface and the level of the tumor cavity would be easy to find and peel . Carbetocin functions as an agonist at peripheral Oxytocin receptors, particularly in the myometrium, resulting in rhythmic contractions of the uterus, increased frequency of existing contractions, and increased uterine tone Terlipressin (triglycyl-lysine vasopressin) became popular in the early 1990s because it has a prolonged duration of action. It is a prodrug and is converted to the lysine vasopressin in the circulation after the N-triglycyl residue is cleaved by endothelial peptidases. This results in a 'slow release' of the vasoactive lysine vasopressin . The effect half-life of terlipressin is 6hr. It causes a prolonged reduction of portal venous pressure (mean 103 min) . The elimination half-life of terlipressin is 50 min .

Owing to its pronounced vasoconstrictive effect within the splanchnic circulation, terlipressin is widely used to treat patients suffering from variceal bleeding during the treatment of hepatorenal syndrome and catecholamine-unresponsive septic shock. Because previous studies have shown a reduction of intravasation by vasopressin during hysteroscopy, we think that its analog, terlipressin, should have the same effect. Terlipressin is an authorized and licensed product used by many clinicians, and its efficacy is supported by sufficient published evidence .

Our study aims to evaluate the efficacy of intramyometrial injection of Terlipressin versus intramyometrial injection of Carbetocin on hemoglobin level in women undergoing abdominal myomectomy. Moreover, to evaluate their efficacy in decreasing blood loss on operative time and to describe the injection sequelae for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 16-45 years
2. Appropriate medical status for laparoscopic surgery (largest myoma ≤15 cm)
3. Baseline hemoglobin ≥9 g/dl
4. No contra-indications to the use of glyopressin or carbitocin
5. Myoma-related symptoms, such as pelvic pressure or pain, menorrhagia, or infertility
6. Not pregnant at the time of presentation (i.e., negative urine pregnancy test or last menstrual period within the last 4 weeks)

Exclusion Criteria:

1. Previous myomectomy
2. History of bleeding disorders
3. Concurrent anticoagulation therapy
4. History of Uncontrolled ischaemic heart disease
5. Any pelvic abnormalities requiring concomitant surgery
6. Treatment with a GnRH agonist or ulipristal acetate within three months preceding surgery
7. Inability to understand and provide written informed consent.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 99 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
effect of intramyometrial terlipressin vs carbitocin vs saline on decreasing blood loss in laparoscopic myomectomy | 12 hours
  1- To evaluate the efficacy of intramyometrial injection of Terlipressin versus intramyometrial injection of Carbetocin in decreasing blood loss in women undergoing laparoscopic myomectomy

SECONDARY OUTCOMES:
effect of intramyometrial terlipressin vs carbitocin vs saline on decrease hemoglobin level in laparoscopic myomectomy | 24 hours
  To evaluate the efficacy of intramyometrial injection of Terlipressin versus intramyometrial injection of Carbetocin on hemoglobin level in women undergoing laparoscopic myomectomy
effect of intramyometrial terlipressin vs carbitocin vs saline on operative time | 12 hours
  2. To evaluate the efficacy of intramyometrial injection of Terlipressin versus intramyometrial injection of Carbetocin on operative time in women undergoing laparoscopic myomectomy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - National Research center, Cairo
  - Wael El Banna Clinic, Maadi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://www.ijrcog.org/index.php/ijrcog/article/view/3925
- Available data/document: Study Protocol — https://ebwhj.journals.ekb.eg/article_125772.html